CLINICAL TRIAL: NCT01956227
Title: Fall Risk Reduction in Multiple Sclerosis: Exercise Versus Behavior
Acronym: FARMS-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMSS-IL-006
Record Dates: First submitted 2013-04-17; First posted 2013-10-08 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis; Adult Disease
MeSH Terms: conditions — Multiple Sclerosis; Disease | interventions — Educational Status; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Home-based Exercise (Experimental): Participants will be taught a series of exercises targeting balance and lower limb strength in four instructional sessions. They will be asked to complete exercises 3 times a week for 12 weeks. Exercise compliance will be recorded with a diary.
  Interventions: Behavioral: Home-based exercise
- Education (Experimental): Participants will attend 4 education sessions focusing on interaction of beliefs, behaviors and symptoms on falls. They will be taught self-management principles to modify their fall risk.
  Interventions: Behavioral: Education
- Exercise plus education (Experimental): Participants will attend 2 instructional exercise sessions as well as 2 education sessions. Participants will be asked to complete exercises at home 3 times per week and engage in behavior to minimize fall risk.
  Interventions: Behavioral: Exercise plus Education
- Control (No Intervention): Participants will not receive any treatment.

INTERVENTIONS:
Behavioral: Home-based exercise — exercise to look at balance and lower limb strength record in diary
  Arms: Home-based Exercise
Behavioral: Education — sessions to discuss self-management ideas to modify risk of falling
  Arms: Education
Behavioral: Exercise plus Education — combination of exercise sessions with education sessions to modify fall risk
  Arms: Exercise plus education

SUMMARY:
Falls are a serious health concern for persons with multiple sclerosis (MS). Over 50% of persons with MS suffer a fall over a 6-month periodwith the majority of falls resulting in medical attention for injuries (i.e., lacerations, bone fractures, & head injuries). The effects of a fall are often compounded as it can lead to activity curtailment, physiological deconditioning, and institutionalization. Despite the importance of falls in persons with MS, the appropriate prevention strategies (i.e. rehabilitation approaches) are not clear. The purpose of this investigation is to determine whether exercise based or educational based interventions are more suited for fall prevention in older adults with MS.

DETAILED DESCRIPTION:
Falls are a serious health concern for persons with multiple sclerosis (MS). Over 50% of persons with MS suffer a fall over a 6-month periodwith the majority of falls resulting in medical attention for injuries (i.e., lacerations, bone fractures, & head injuries). The effects of a fall are often compounded as it can lead to activity curtailment, physiological deconditioning, and institutionalization. Despite the importance of falls in persons with MS, the appropriate prevention strategies (i.e. rehabilitation approaches) are not clear.

It is well known that causes of falls are multifactorial with over 400 risk factors identified. However, it is believed that these factors can be divided into two main classes: intrinsic (e.g. physiological factors) and extrinsic factors. For instance balance dysfunction, spasticity and muscle weakness are physiological risk factors for falls in MS . Behavioral fall risk factors in MS include choosing appropriate footwear, lighting and utilizing appropriate assistive device. There is evidence that both types of risk factors can be minimized with appropriately designed interventions in persons with MS and have been shown to reduce fall risk and incidence in other clinical populations. This has led to calls for the combination of exercise training program that targets specific, modifiable physiological risk factors and educational interventions targeting modifiable behavioral risk factors in persons with MS. However, there is minimal evidence that these interventions in isolation or combination actually reduce fall incidence or risk in persons with MS. This proposal seeks to determine the effectiveness of a combined exercise and educational rehabilitation strategy to prevent falls in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* Definite multiple sclerosis diagnosis
* ambulatory
* aged 50-75 years of age
* fallen within 12 months

Exclusion Criteria:

* non-ambulatory
* outside age range
* no fall history

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Fall incidence | 3 months

SECONDARY OUTCOMES:
Physiological Fall Risk | 3 Months
  Physiological fall risk will be determined by the short form of the Physiological Profile Assessment (PPA)(Lord, 2003). The PPA is a standardized test battery which assesses vision (edge contrast sensitivity), lower limb proprioception, strength (knee extension), postural sway, and cognitive function (simple hand reaction time). The outcome of each test will be combined to generate an overall fall risk score
Mobility | 3 months
  Specific measures of walking speed, endurance, coordination and self-reported walking function scale will be employed to assess overall mobility of each person. Walking speed was quantified with the Timed 25-Foot Walk (T25W), walking endurance was assessed with the 6-Minute Walk (6MW), and functional mobility was quantified with the Timed Up and Go (TUG) . The Multiple Sclerosis Walking Scale-12 (MSWS-12) will be used as a self-reported measure of walking impairment.
Balance | 3 Months
  To assess balance (e.g. postural control), we conducted a clinical assessment To measure balance the Berg Balance Scale (BBS) and self-reports of balance confidence will be used. The BBS is a clinical assessment of balance. Scores on the BBS range from 0-56 with higher scores indicating greater balance. The Activities-Specific Balance Confidence (ABC) scale was used as a measure of balance confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sosnoff, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois UC, Urbana, Illinois, United States

REFERENCES:
- [Derived] Sosnoff JJ, Moon Y, Wajda DA, Finlayson ML, McAuley E, Peterson EW, Morrison S, Motl RW. Fall risk and incidence reduction in high risk individuals with multiple sclerosis: a pilot randomized control trial. Clin Rehabil. 2015 Oct;29(10):952-60. doi: 10.1177/0269215514564899. Epub 2014 Dec 23. PMID 25540170